CLINICAL TRIAL: NCT02898207
Title: A Phase 1 Study of PARP Inhibitor Olaparib and HSP90 Inhibitor AT13387 for Treatment of Advanced Solid Tumors With Expansion in Patients With Recurrent Epithelial Ovarian, Fallopian Tube, Peritoneal Cancer or Recurrent Triple-Negative Breast Cancer
Brief Title: Olaparib and Onalespib in Treating Patients With Solid Tumors That Are Metastatic or Cannot Be Removed by Surgery or Recurrent Ovarian, Fallopian Tube, Primary Peritoneal, or Triple-Negative Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2016-01364; NCI-2016-01364 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 17-715; 10031 (Other: Dana-Farber - Harvard Cancer Center LAO); 10031 (Other: CTEP); UM1CA186709 (NIH)
Record Dates: First submitted 2016-09-12; First posted 2016-09-13 (Estimated); Results first posted 2023-04-26 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Metastatic High Grade Fallopian Tube Serous Adenocarcinoma; Metastatic Malignant Solid Neoplasm; Metastatic Primary Peritoneal Serous Adenocarcinoma; Metastatic Triple-Negative Breast Carcinoma; Platinum-Resistant Fallopian Tube Carcinoma; Platinum-Resistant Ovarian Carcinoma; Platinum-Resistant Primary Peritoneal Carcinoma; Recurrent Breast Carcinoma; Recurrent High Grade Fallopian Tube Serous Adenocarcinoma; Recurrent High Grade Ovarian Serous Adenocarcinoma; Recurrent Primary Peritoneal High Grade Serous Adenocarcinoma; Recurrent Triple-Negative Breast Carcinoma; Refractory Fallopian Tube Serous Adenocarcinoma; Refractory Ovarian Serous Adenocarcinoma; Refractory Primary Peritoneal Serous Adenocarcinoma; Refractory Triple-Negative Breast Carcinoma; Unresectable High Grade Fallopian Tube Serous Adenocarcinoma; Unresectable Malignant Solid Neoplasm; Unresectable Primary Peritoneal Serous Adenocarcinoma
MeSH Terms: conditions — Neoplasm Metastasis; Triple Negative Breast Neoplasms; Breast Neoplasms | interventions — olaparib; (2,4-dihydroxy-5-isopropylphenyl)-(5-(4-methylpiperazin-1-ylmethyl)-1,3-dihydroisoindol-2-yl)methanone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Dose Level 0: Olaparib 200 mg and Onalespib 20 mg/m^2 (Experimental): Dose Level 0 (DL0): Patients received olaparib 200 mg PO BID on days 1-7 (cycle 0). Beginning in cycle 1, patients received olaparib 200mg PO BID on days 1-28 and onalespib 20 mg/m^2 IV over 1 hour on days 1, 2, 8, 9, 15, and 16. Cycles repeated every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Olaparib; Drug: Onalespib
- Dose Level 1: Olaparib 200 mg and Onalespib 40 mg/m^2 (Experimental): Dose Level 1 (DL1): Patients received olaparib 200 mg PO BID on days 1-7 (cycle 0). Beginning in cycle 1, patients received olaparib 200mg PO BID on days 1-28 and onalespib 40 mg/m^2 IV over 1 hour on days 1, 2, 8, 9, 15, and 16. Cycles repeated every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Olaparib; Drug: Onalespib
- Dose Level 2: Olaparib 300 mg and Onalespib 40 mg/m^2 (Experimental): Dose Level 2 (DL2): Patients received olaparib 300 mg PO BID on days 1-7 (cycle 0). Beginning in cycle 1, patients received olaparib 300 mg PO BID on days 1-28 and onalespib 40 mg/m^2 IV over 1 hour on days 1, 2, 8, 9, 15, and 16. Cycles repeated every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Olaparib; Drug: Onalespib
- Dose Level 3: Olaparib 300 mg and Onalespib 80 mg/m^2 (Experimental): Dose Level 3 (DL3): Patients received olaparib 300 mg PO BID on days 1-7 (cycle 0). Beginning in cycle 1, patients received olaparib 300 mg PO BID on days 1-28 and onalespib 80 mg/m^2 IV over 1 hour on days 1, 2, 8, 9, 15, and 16. Cycles repeated every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Olaparib; Drug: Onalespib
- Dose Level 2a: Olaparib 200 mg and Onalespib 80 mg/m^2 (Experimental): Dose Level 2a (DL2a): Patients received olaparib 200 mg PO BID on days 1-7 (cycle 0). Beginning in cycle 1, patients received olaparib 200 mg PO BID on days 1-28 and onalespib 80 mg/m^2 IV over 1 hour on days 1, 2, 8, 9, 15, and 16. Cycles repeated every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Olaparib; Drug: Onalespib
- Dose Level 3a: Olaparib 200 mg and Onalespib 120 mg/m^2 (Experimental): Dose Level 3a (DL3a): Patients received olaparib 200 mg PO BID on days 1-7 (cycle 0). Beginning in cycle 1, patients received olaparib 200 mg PO BID on days 1-28 and onalespib 120 mg/m^2 IV over 1 hour on days 1, 2, 8, 9, 15, and 16. Cycles repeated every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Olaparib; Drug: Onalespib

INTERVENTIONS:
Drug: Olaparib — Given PO
  Other Names: AZD 2281; AZD-2281; AZD2281; KU-0059436; Lynparza; PARP Inhibitor AZD2281
Drug: Onalespib — Given IV
  Other Names: AT 13387; AT-13387; AT13387

SUMMARY:
This phase I trial studies the side effects and best dose of olaparib and onalespib when given together in treating patients with solid tumors that have spread to other places in the body (metastatic) or cannot be removed by surgery (unresectable) or ovarian, fallopian tube, primary peritoneal, or triple-negative breast cancer that has come back (recurrent). Olaparib and onalespib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To establish the maximum tolerated dose (MTDs) of olaparib and onalespib (AT13387) administered in combination in patients with advanced solid tumors.

SECONDARY OBJECTIVES:

I. To identify the dose-limiting toxicity (DLT) and other toxicities associated with olaparib and AT13387 administered in combination as assessed by Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0.

II. To determine the recommended phase 2 doses (RP2D) of the combination of olaparib and AT13387.

III. To determine the plasma pharmacokinetics of olaparib and AT13387. IV. To document anti-tumor activity of the combination of olaparib and AT13387 as assessed by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and progression free survival (PFS). Although the clinical benefit of [this/these] drug(s) has not yet been established, the intent of offering this treatment is to provide a possible therapeutic benefit, and thus the patient will be carefully monitored for tumor response and symptom relief in addition to safety and tolerability.

OUTLINE: This is a dose-escalation study.

Patients receive olaparib orally (PO) twice daily (BID) on days 1-7 (cycle 0). Beginning in cycle 1, patients receive olaparib PO BID on days 1-28 and onalespib intravenously (IV) over 1 hour on days 1, 2, 8, 9, 15, and 16. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and every 3 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* For the dose escalation cohort, patients must have histologically or cytologically confirmed malignancy that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective
* For the dose escalation cohort, patients may have received any number of prior therapies
* For the dose expansion cohort, participants must have histologically or cytologically confirmed diagnosis of either:

  * Ovarian, fallopian tube, or primary peritoneal cancer of high grade serous histology which has recurred despite standard therapy; up to 3 prior lines in the platinum resistant setting (i.e. up to 3 lines after patients have become platinum resistant); patients may have received unlimited lines while platinum sensitive
  * Triple-negative breast cancer (TNBC) which has recurred despite standard therapy; recurrent TNBC needs to have metastatic disease and patients with an in breast recurrence are not eligible; up to 4 prior lines in the recurrent setting for patients with triple-negative breast cancer are allowed
* For the dose expansion cohort, patients with ovarian, fallopian tube or primary peritoneal cancer must have platinum resistant disease defined as progression within 6 months after last platinum regimen; platinum refractory disease is allowed
* For the dose expansion cohort, patients with triple-negative breast cancer may not be BRCA1/2 germline mutation carriers
* Because no dosing or adverse event data are currently available on the use of olaparib in combination with AT13387 in patients < 18 years of age, children are excluded from this study, but will be eligible for future pediatric trials.
* There must be availability of a formalin-fixed, paraffin-embedded tumor specimen
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 (Karnofsky > 60%)
* Life expectancy of greater than 12 weeks
* Leukocytes >= 3,000/mcL
* Hemoglobin >= 10 g/dL with no blood transfusion in the past 28 days
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x institutional upper limit of normal
* Creatinine =< the institutional upper limit of normal OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Corrected QT using Fridericia's formula (QTcF) =< 450 ms
* Any clinically significant electrolyte imbalance, particularly hypokalemia and hypomagnesemia, should be corrected before treatment
* Pre-study evaluation must include an ophthalmologic exam by an ophthalmologist (not optometrist) and should minimally include visual acuity testing, slit lamp examination, and funduscopic examination; follow up eye-exams will only be performed if subjects develop/report any visual impairment; visual impairment may include peripheral flashes (photopsia), blurred or double vision, floaters, color distortion and dimness, difficulties with light/dark accommodation, tunnel vision or other field defects, halos, apparent movement of stationary objects, and complex disturbances; follow up eye-exams will minimally include visual acuity testing, slit lamp examination, and funduscopic examination; additional testing will be based on symptoms, what is observed and ophthalmologist recommendations
* For the expansion cohort only: measurable disease by RECIST v1.1 with at least one measurable target lesion
* The effects of olaparib in combination with AT13387on the developing human fetus are unknown; for this reason and because olaparib and AT13387 are anti-neoplastic small molecule inhibitors, which are agents that are potentially teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 3 months after the last dose of study drugs; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of olaparib and/or AT13387 administration
* Patients must be able to swallow tablets and have no significant impairment in gastrointestinal absorption
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* All acute, clinically significant treatment-related toxicity from prior therapy, except for alopecia, must have resolved to grade =< 1
* Patients who are receiving any other investigational agents
* Patients with known active or history of brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to olaparib and AT13387 used in study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because olaparib and AT13387 are agents with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with AT13387 or olaparib, breastfeeding should be discontinued if the mother is treated with olaparib or AT13387
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with olaparib or AT13387; in addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated
* Known history of QT/corrected QT (QTc) prolongation or torsades de pointes (TdP); patients who are currently receiving treatment with medication with a known risk to prolong the QT interval or inducing torsades de pointes and the treatment cannot either be discontinued or switched to a different medication prior to starting study drugs
* Participants receiving any medications or substances that are strong inhibitors or inducers of CYP3A4 or moderate inhibitors of CYP3A4 are ineligible; the study team should check a frequently-updated medical reference for a list of drugs to avoid or minimize use of; as part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Participants with myelodysplastic syndrome/acute myeloid leukemia or with features suggestive of myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-05-19 (Actual); Primary Completion 2020-07-29 (Actual); Study Completion 2022-01-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Panagiotis A Konstantinopoulos, Principal Investigator — Dana-Farber - Harvard Cancer Center LAO
Locations (8):
- United States (8):
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic in Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Dose Level 0
Arm/Group | Dose Level 0: Olaparib 200 mg and Onalespib 20 mg/m^2 | Dose Level 1: Olaparib 200 mg and Onalespib 40 mg/m^2 | Dose Level 2: Olaparib 300 mg and Onalespib 40 mg/m^2 | Dose Level 3: Olaparib 300 mg and Onalespib 80 mg/m^2 | Dose Level 2a: Olaparib 200 mg and Onalespib 80 mg/m^2 | Dose Level 3a: Olaparib 200 mg and Onalespib 120 mg/m^2
Started | 3 | 0 | 0 | 0 | 0 | 0
Completed | 3 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Dose Level 1
Arm/Group | Dose Level 0: Olaparib 200 mg and Onalespib 20 mg/m^2 | Dose Level 1: Olaparib 200 mg and Onalespib 40 mg/m^2 | Dose Level 2: Olaparib 300 mg and Onalespib 40 mg/m^2 | Dose Level 3: Olaparib 300 mg and Onalespib 80 mg/m^2 | Dose Level 2a: Olaparib 200 mg and Onalespib 80 mg/m^2 | Dose Level 3a: Olaparib 200 mg and Onalespib 120 mg/m^2
Started | 0 | 4 | 0 | 0 | 0 | 0
Completed | 0 | 4 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Dose Level 2
Arm/Group | Dose Level 0: Olaparib 200 mg and Onalespib 20 mg/m^2 | Dose Level 1: Olaparib 200 mg and Onalespib 40 mg/m^2 | Dose Level 2: Olaparib 300 mg and Onalespib 40 mg/m^2 | Dose Level 3: Olaparib 300 mg and Onalespib 80 mg/m^2 | Dose Level 2a: Olaparib 200 mg and Onalespib 80 mg/m^2 | Dose Level 3a: Olaparib 200 mg and Onalespib 120 mg/m^2
Started | 0 | 0 | 6 | 0 | 0 | 0
Completed | 0 | 0 | 6 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Dose Level 3
Arm/Group | Dose Level 0: Olaparib 200 mg and Onalespib 20 mg/m^2 | Dose Level 1: Olaparib 200 mg and Onalespib 40 mg/m^2 | Dose Level 2: Olaparib 300 mg and Onalespib 40 mg/m^2 | Dose Level 3: Olaparib 300 mg and Onalespib 80 mg/m^2 | Dose Level 2a: Olaparib 200 mg and Onalespib 80 mg/m^2 | Dose Level 3a: Olaparib 200 mg and Onalespib 120 mg/m^2
Started | 0 | 0 | 0 | 7 | 0 | 0
Completed | 0 | 0 | 0 | 7 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Dose Level 2a
Arm/Group | Dose Level 0: Olaparib 200 mg and Onalespib 20 mg/m^2 | Dose Level 1: Olaparib 200 mg and Onalespib 40 mg/m^2 | Dose Level 2: Olaparib 300 mg and Onalespib 40 mg/m^2 | Dose Level 3: Olaparib 300 mg and Onalespib 80 mg/m^2 | Dose Level 2a: Olaparib 200 mg and Onalespib 80 mg/m^2 | Dose Level 3a: Olaparib 200 mg and Onalespib 120 mg/m^2
Started | 0 | 0 | 0 | 0 | 3 | 0
Completed | 0 | 0 | 0 | 0 | 3 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Dose Level 3a
Arm/Group | Dose Level 0: Olaparib 200 mg and Onalespib 20 mg/m^2 | Dose Level 1: Olaparib 200 mg and Onalespib 40 mg/m^2 | Dose Level 2: Olaparib 300 mg and Onalespib 40 mg/m^2 | Dose Level 3: Olaparib 300 mg and Onalespib 80 mg/m^2 | Dose Level 2a: Olaparib 200 mg and Onalespib 80 mg/m^2 | Dose Level 3a: Olaparib 200 mg and Onalespib 120 mg/m^2
Started | 0 | 0 | 0 | 0 | 0 | 5
Completed | 0 | 0 | 0 | 0 | 0 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 0: Olaparib 200 mg and Onalespib 20 mg/m^2 | Dose Level 1: Olaparib 200 mg and Onalespib 40 mg/m^2 | Dose Level 2: Olaparib 300 mg and Onalespib 40 mg/m^2 | Dose Level 3: Olaparib 300 mg and Onalespib 80 mg/m^2 | Dose Level 2a: Olaparib 200 mg and Onalespib 80 mg/m^2 | Dose Level 3a: Olaparib 200 mg and Onalespib 120 mg/m^2 | Total
Number analyzed (Participants) | 3 | 4 | 6 | 7 | 3 | 5 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (11.6) | 60.8 (8.5) | 59.8 (10.6) | 57 (11.1) | 66.7 (1.2) | 65.4 (5.9) | 61.5 (9.2)
Age, Continuous [Median (Full Range); unit: years] | 59 [57 to 78] | 65 [48 to 65] | 57.5 [45 to 76] | 53 [46 to 72] | 66 [66 to 68] | 66 [56 to 72] | 65 [45 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 5 | 6 | 3 | 5 | 26
  Male | 0 | 0 | 1 | 1 | 0 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 4 | 6 | 7 | 3 | 5 | 28
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 3 | 2 | 6 | 6 | 3 | 5 | 25
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 3 | 4 | 6 | 7 | 3 | 5 | 28
ECOG Performance Status [Count of Participants; unit: Participants]
  0 = Asymptomatic and fully active | 1 | 4 | 2 | 4 | 2 | 4 | 17
  1 = Symptomatic; fully ambulatory; restricted in physically strenuous activity | 2 | 0 | 4 | 3 | 1 | 1 | 11
Primary Site of Disease [Count of Participants; unit: Participants]
  Ovary | 3 | 2 | 2 | 5 | 3 | 3 | 18
  Uterus | 0 | 2 | 1 | 0 | 0 | 2 | 5
  Colon | 0 | 0 | 1 | 1 | 0 | 0 | 2
  Breast | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Melanoma | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Malignant solitary fibrous tumor | 0 | 0 | 1 | 0 | 0 | 0 | 1
Stage at Diagnosis [Count of Participants; unit: Participants] — Measure Description: Staging was based on the FIGO (International Federation of Gynecology and Obstetrics) and AJCC (American Joint Committee on Cancer) systems. Stage I cancers usually have not grown deeply into nearby tissues. Stage II and III cancers have grown more deeply into nearby tissue and may have spread to lymph nodes. Stage IV cancers have spread to other organs or parts of the body. Higher stages are typically associated with worse outcomes.
  Participants
    IC | 0 | 0 | 0 | 0 | 0 | 1 | 1
    IIC | 0 | 0 | 0 | 0 | 1 | 0 | 1
    III | 1 | 1 | 0 | 1 | 0 | 0 | 3
    IIIC | 0 | 2 | 2 | 0 | 0 | 1 | 5
    IV | 2 | 1 | 4 | 5 | 2 | 0 | 14
    IVB | 0 | 0 | 0 | 1 | 0 | 3 | 4
Histology [Count of Participants; unit: Participants]
  Well differentiated | 0 | 1 | 1 | 0 | 0 | 0 | 2
  Moderately differentiated | 1 | 0 | 1 | 0 | 0 | 0 | 2
  Poorly differentiated | 0 | 3 | 2 | 4 | 2 | 4 | 15
  Grade cannot be assessed/unknown | 2 | 0 | 2 | 3 | 1 | 1 | 9
Lines of Prior Therapy [Median (Full Range); unit: Lines of prior therapy] | 5 [3 to 11] | 3 [2 to 7] | 5.5 [2 to 15] | 6 [4 to 12] | 7 [6 to 11] | 3 [1 to 8] | 5.5 [1 to 15]

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Olaparib Administered in Combination With Onalespib
Description: MTD was determined by testing increasing doses of the combination of olaparib PO and onalespib IV within dose escalation cohorts consisting of 3 to 6 evaluable participants. MTD reflects the highest dose combination that did not cause a Dose-Limiting Toxicity (DLT) in > 33% of participants. DLTs were defined based on the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0.
  Enrollment to this study was suspended prior to completion of the dose escalation due to discontinuation of further development of onalespib. A true single MTD therefore could not be determined. The two dose levels included in this outcome measure represent the highest well-tolerated dose combinations (Dose Level 2 [DL2]: Olaparib 300 mg PO BID and Onalespib 40 mg/m^2 IV; and Dose Level 2a [DL2a]: Olaparib 200 mg PO BID and Onalespib 80 mg/m^2 IV).
Time Frame: Up to 35 days for each dose level cohort
Population: Seven of the 28 patients were not evaluable for DLT assessment and were replaced.
Measure: Number; unit: mg
Groups:
- All Evaluable Participants: All participants who received at least 75% of planned olaparib and at least 4 doses of onalespib within the DLT period.
Arm/Group | All Evaluable Participants
Number analyzed (Participants) | 21
mg
  Dose Level 2 Olaparib PO BID | 300
  Dose Level 2a Olaparib PO BID | 200

2. Primary Outcome: Maximum Tolerated Dose (MTD) of Onalespib Administered in Combination With Olaparib
Description: MTD was determined by testing increasing doses of the combination of olaparib PO and onalespib IV within dose escalation cohorts consisting of 3 to 6 evaluable participants. MTD reflects the highest dose combination that did not cause a Dose-Limiting Toxicity (DLT) in > 33% of participants. DLTs were defined based on the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0.
Time Frame: Up to 35 days for each dose level cohort
Population: Seven of the 28 patients were not evaluable for DLT assessment and were replaced.
Measure: Number; unit: mg/m2
Arm/Group | All Evaluable Participants
Number analyzed (Participants) | 21
mg/m2
  Dose Level 2 Onalespib IV on Days 1, 2, 8, 9, 15, and 16 | 40
  Dose Level 2a Onalespib IV on Days 1, 2, 8, 9, 15, and 16 | 80

3. Secondary Outcome: Number of Participants Who Experienced Dose-Limiting Toxicities (DLTs)
Description: DLTs were based on the NCI Common Terminology Criteria for Adverse Events (CTCAE) v.5.0 and were defined as any grade 3 or 4 non-hematologic toxicity (excluding grade 3: fatigue; diarrhea, constipation, and nausea and/or vomiting controlled with supportive measured within 24 hours; hypophosphatemia; hyponatremia; hypomagnesemia; and rash that resolves to < grade 3 within < 5 days), grade 4 neutropenia of > 7 day duration, febrile neutropenia, grade 4 thrombocytopenia or bleeding associated with grade 3 thrombocytopenia, requirement for repeated blood transfusion within 4-6 weeks, any other grade 4 hematologic toxicity, any study treatment-related death, any grade 3 or 4 event considered to be dose-limiting in the opinion of the investigator, and the inability to take 75% or more of the planned dose for olaparib and 4 out of 6 doses for onalespib within the DLT period due to treatment-related adverse events.
Time Frame: Within Cycles 0 and 1 (up to 35 days).
Population: Patients were considered not evaluable for the DLT outcome if they did not receive at least 75% of the planned olaparib doses or at least 4 doses of onalespib for reasons other than toxicity or DLT. Dose Level 3a did not complete evaluation as enrollment was suspended due to discontinuation of further development of onalespib.
Measure: Count of Participants; unit: Participants
Groups:
- Dose Level 3: Olaparib 300 mg and Onalespib 80 mg/m^: Dose Level 3 (DL3): Patients received olaparib 300 mg PO BID on days 1-7 (cycle 0). Beginning in cycle 1, patients received olaparib 300 mg PO BID on days 1-28 and onalespib 80 mg/m^2 IV over 1 hour on days 1, 2, 8, 9, 15, and 16. Cycles repeated every 28 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | Dose Level 0: Olaparib 200 mg and Onalespib 20 mg/m^2 | Dose Level 1: Olaparib 200 mg and Onalespib 40 mg/m^2 | Dose Level 2: Olaparib 300 mg and Onalespib 40 mg/m^2 | Dose Level 3: Olaparib 300 mg and Onalespib 80 mg/m^ | Dose Level 2a: Olaparib 200 mg and Onalespib 80 mg/m^2 | Dose Level 3a: Olaparib 200 mg and Onalespib 120 mg/m^2
Number analyzed (Participants) | 3 | 3 | 3 | 5 | 3 | 4
Participants | 0 | 0 | 0 | 0 | 2 | 1

4. Secondary Outcome: Number of Participants Who Experienced Treatment-Related Toxicities
Description: Treatment-related toxicities in this outcome include non-hematologic and hematologic adverse events that were either Grade 3+ or occurred in at least 10% of all treated participants, and were considered at least possibly related to olaparib and/or onalespib. Adverse events were graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) v.5.0.
Time Frame: Up to 67 weeks
Population: One patient was enrolled under Dose Level 3, but was erroneously treated at Dose Level 2. This patient was replaced within the dose escalation, but remained on treatment on Dose Level 2 throughout the remainder of trial participation. For the purposes of adverse event reporting, this patient has been included in Dose Level 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 0: Olaparib 200 mg and Onalespib 20 mg/m^2 | Dose Level 1: Olaparib 200 mg and Onalespib 40 mg/m^2 | Dose Level 2: Olaparib 300 mg and Onalespib 40 mg/m^2 | Dose Level 3: Olaparib 300 mg and Onalespib 80 mg/m^2 | Dose Level 2a: Olaparib 200 mg and Onalespib 80 mg/m^2 | Dose Level 3a: Olaparib 200 mg and Onalespib 120 mg/m^2
Number analyzed (Participants) | 3 | 4 | 7 | 6 | 3 | 5
Participants
  Diarrhea : Maximum Grade 1-2 | 3 | 3 | 3 | 5 | 3 | 4
  Diarrhea : Maximum Grade 3 | 0 | 0 | 0 | 0 | 0 | 1
  Nausea : Maximum Grade 1-2 | 1 | 2 | 4 | 6 | 3 | 2
  Nausea : Maximum Grade 3 | 1 | 0 | 0 | 0 | 0 | 0
  Anemia : Maximum Grade 1-2 | 2 | 3 | 2 | 4 | 1 | 1
  Anemia : Maximum Grade 3 | 0 | 0 | 0 | 2 | 0 | 3
  Thrombocytopenia/platelet count decrease : Maximum Grade 1-2 | 0 | 3 | 1 | 3 | 0 | 3
  Thrombocytopenia/platelet count decrease : Maximum Grade 3 | 0 | 0 | 0 | 1 | 0 | 1
  Fatigue : Maximum Grade 1-2 | 1 | 3 | 3 | 2 | 1 | 2
  Vomiting : Maximum Grade 1-2 | 1 | 1 | 3 | 2 | 1 | 0
  Vomiting : Maximum Grade 3 | 1 | 0 | 0 | 0 | 0 | 0
  Abdominal pain : Maximum Grade 1-2 | 1 | 1 | 0 | 0 | 2 | 0
  Abdominal pain : Maximum Grade 3 | 0 | 0 | 1 | 0 | 0 | 0
  Anorexia : Maximum Grade 1-2 | 1 | 1 | 1 | 0 | 1 | 1
  Neutrophil count decreased : Maximum Grade 1-2 | 0 | 0 | 1 | 1 | 0 | 1
  Neutrophil count decreased : Maximum Grade 4 | 0 | 0 | 0 | 0 | 0 | 1
  Lymphocyte count decreased : Maximum Grade 1-2 | 0 | 0 | 0 | 1 | 1 | 1
  Lymphocyte count decreased : Maximum Grade 3 | 0 | 0 | 0 | 0 | 0 | 1
  Floaters : Maximum Grade 1-2 | 0 | 1 | 0 | 1 | 0 | 2
  Dysgeusia : Maximum Grade 1-2 | 0 | 1 | 0 | 1 | 0 | 2

5. Secondary Outcome: Number of Participants With Objective Responses by RECIST 1.1
Description: Responses determined per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by CT or MRI, where Objective Response (OR) represents either a Complete Response (CR; disappearance of all target lesions) or a Partial Response (PR; at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum diameters).
Time Frame: Up to 63 weeks
Population: Only participants who had their disease re-evaluated via CT or MRI were considered evaluable for response. Six of the 28 participants were taken off study therapy prior to their first on-study disease evaluation.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 0: Olaparib 200 mg and Onalespib 20 mg/m^2 | Dose Level 1: Olaparib 200 mg and Onalespib 40 mg/m^2 | Dose Level 2: Olaparib 300 mg and Onalespib 40 mg/m^2 | Dose Level 3: Olaparib 300 mg and Onalespib 80 mg/m^2 | Dose Level 2a: Olaparib 200 mg and Onalespib 80 mg/m^2 | Dose Level 3a: Olaparib 200 mg and Onalespib 120 mg/m^2
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 4
Participants | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants Progression-Free for At Least 24 Weeks by RECIST 1.1
Description: Responses determined per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by CT or MRI, where Progressive Disease (PD) represents (relative to baseline) at least a 20% increase in the sum of diameters of target lesions, appearance of one or more new lesions, or unequivocal progression of existing non-target lesions. The duration of progression-free status was defined as the interval from the date of enrollment to date of either PD or date of last disease assessment.
Time Frame: Up to 24 weeks
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 0: Olaparib 200 mg and Onalespib 20 mg/m^2 | Dose Level 1: Olaparib 200 mg and Onalespib 40 mg/m^2 | Dose Level 2: Olaparib 300 mg and Onalespib 40 mg/m^2 | Dose Level 3: Olaparib 300 mg and Onalespib 80 mg/m^2 | Dose Level 2a: Olaparib 200 mg and Onalespib 80 mg/m^2 | Dose Level 3a: Olaparib 200 mg and Onalespib 120 mg/m^2
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 4
Participants | 1 | 2 | 1 | 1 | 1 | 1

ADVERSE EVENTS:
Time Frame: Adverse events data was collected throughout study participation for all patients from first administration through 30 days of the last administration of the investigational agent(s), up to 67 weeks.
Description: One patient was enrolled under Dose Level 3, but was erroneously treated at Dose Level 2. This patient was replaced within the dose escalation, but remained on treatment on Dose Level 2 throughout the remainder of trial participation. For the purposes of adverse event reporting, this patient has been included in Dose Level 2.
Groups:
- Dose Level 0: Cycle 0 Dose: Olaparib 200 mg PO BID; Cycle 1+ Dose: Olaparib 200 mg PO BID, Onalespib 20 mg/m2 IV on days 1, 2, 8, 9, 15, and 16
- Dose Level 1: Cycle 0 Dose: Olaparib 200 mg PO BID; Cycle 1+ Dose: Olaparib 200 mg PO BID, Onalespib 40 mg/m2 IV on days 1, 2, 8, 9, 15, and 16
- Dose Level 2: Cycle 0 Dose: Olaparib 300 mg PO BID; Cycle 1+ Dose: Olaparib 300 mg PO BID, Onalespib 40 mg/m2 IV on days 1, 2, 8, 9, 15, and 16
- Dose Level 3: Cycle 0 Dose: Olaparib 300 mg PO BID; Cycle 1+ Dose: Olaparib 300 mg PO BID, Onalespib 80 mg/m2 IV on days 1, 2, 8, 9, 15, and 16
- Dose Level 2a: Cycle 0 Dose: Olaparib 200 mg PO BID; Cycle 1+ Dose: Olaparib 200 mg PO BID, Onalespib 80 mg/m2 IV on days 1, 2, 8, 9, 15, and 16
- Dose Level 3a: Cycle 0 Dose: Olaparib 200 mg PO BID; Cycle 1+ Dose: Olaparib 200 mg PO BID, Onalespib 120 mg/m2 IV on days 1, 2, 8, 9, 15, and 16
Arm/Group | Dose Level 0 | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 2a | Dose Level 3a
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4 | 0/7 | 1/6 | 0/3 | 0/5
Serious Adverse Events (participants affected / at risk) | 2/3 | 2/4 | 4/7 | 2/6 | 0/3 | 2/5
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 7/7 | 6/6 | 3/3 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 0 (N=3) | Dose Level 1 (N=4) | Dose Level 2 (N=7) | Dose Level 3 (N=6) | Dose Level 2a (N=3) | Dose Level 3a (N=5)
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pericardial tamponade (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
General and admin site - Other - Disease Progression (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Colonic obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 0 | 0
Rectal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0 | 0
Small intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nervous system - Other - Brain Mets (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Resp, thoracic & mediast - Other - Pulmonary Embous (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 0 (N=3) | Dose Level 1 (N=4) | Dose Level 2 (N=7) | Dose Level 3 (N=6) | Dose Level 2a (N=3) | Dose Level 3a (N=5)
Diarrhea (Gastrointestinal disorders) | 3 | 3 | 4 | 4 | 3 | 5
Nausea (Gastrointestinal disorders) | 2 | 3 | 6 | 6 | 3 | 2
Anemia (Blood and lymphatic system disorders) | 2 | 3 | 5 | 5 | 2 | 4
Fatigue (General disorders) | 2 | 3 | 4 | 3 | 1 | 2
Vomiting (Gastrointestinal disorders) | 2 | 2 | 5 | 2 | 1 | 1
Platelet count decreased (Investigations) | 0 | 3 | 1 | 4 | 0 | 4
Abdominal pain (Gastrointestinal disorders) | 2 | 3 | 3 | 1 | 2 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 1 | 3 | 1 | 2 | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 2 | 2 | 3 | 0 | 0
Creatinine increased (Investigations) | 1 | 1 | 2 | 1 | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 2 | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 1 | 2 | 2 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 1 | 2 | 1 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 2 | 0 | 1
Floaters (Eye disorders) | 0 | 1 | 0 | 1 | 1 | 2
Bloating (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1 | 1
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 2
Headache (Nervous system disorders) | 0 | 0 | 1 | 1 | 1 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 1 | 0 | 2
Pain (General disorders) | 1 | 1 | 1 | 0 | 0 | 1
AST increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 1
Alkaline phosphatase increased (Investigations) | 0 | 1 | 1 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 2 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 1
Edema limbs (General disorders) | 1 | 1 | 0 | 0 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 2 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0 | 0
Weight loss (Investigations) | 1 | 0 | 1 | 0 | 0 | 1
ALT increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0
Colonic obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Hot flashes (Vascular disorders) | 1 | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0
Allergic reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Blood/Lymph - Other - Low Iron (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Flashing lights (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal disorders - Other, specify - Belching (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal disorders - Other, specify - Burping/Belching (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
General and admin site - Other - Disease Progression (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
General and admin site - Other - Increased Phelgm (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
General and admin site - Other - Lightheaded (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Infections and infestations - Other - Fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Infections and infestations - Other - Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Infections and infestations - Other - Sinus Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Investigations - Other, specify - Taste Changes (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Lip infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Metabolism and nutrition - Other - Altered Taste (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Musculoskel/connect tissue -Other - Intermittent Muscle Cramps (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Musculoskel/connect tissue -Other - Muscle Cramps (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nervous system disorders - Other - Brain Mets (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nervous system disorders - Other - Night Sweats (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nervous system disorders - Other - Nightmares (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nervous system disorders - Other - Shakiness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Paresthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pericardial tamponade (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rectal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Renal and urinary disorders - Other - Bladder Pressure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Resp, thoracic & mediast - Other - Cold Symptoms (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Resp, thoracic & mediast - Other - Increased Phlegm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Resp, thoracic & mediast - Other - Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Resp, thoracic & mediast - Other - Pulmonary Embous (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Skin & subcutaneous tissue -Other - Night Sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Small intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Spasticity (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Surgical and medical - Other - Colectomy (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Urinary frequency (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Urinary urgency (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
White blood cell decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-10): https://cdn.clinicaltrials.gov/large-docs/07/NCT02898207/Prot_SAP_000.pdf